CLINICAL TRIAL: NCT05999526
Title: Mechanical Ventilation Reconnection for One Hour After Spontaneous Breathing Trial: a Randomized Controlled Feasibility Trial
Brief Title: Mechanical Ventilation Reconnection for One Hour After Spontaneous Breathing Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Hospitalar Unimed de Joinville (Other)
Responsible Party: Principal Investigator, Aline Braz Pereira, Principal Investigator, Centro Hospitalar Unimed de Joinville
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHUnimed; 70984323.1.1001.5362 (Registry Identifier: Certificate of Presentation of Ethical Appreciation)
Record Dates: First submitted 2023-08-12; First posted 2023-08-21 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2024-02

CONDITIONS: Airway Extubation; Ventilator Weaning
Keywords: Rest; Ventilator Weaning; Airway Extubation

STUDY DESIGN:
Intervention Model Description: Immediately after successful spontaneous breathing trial, eligible participants will be randomized into 2 groups that will undergo the following interventions:
  1. Reconnection to mechanical ventilation for 1 hour: as soon as the success of the spontaneous breathing trial is confirmed, the participants will be reconnected to mechanical ventilator for 1 hour using the previous ventilatory parameters and, afterwards, extubated.
     In the experimental group, in case there are signs of respiratory distress or other clinical problems during the resting phase on mechanical ventilation, the intensivist may decide to keep the participant on mechanical ventilation for more than 1 hour until reassessing the appropriate time for extubation.
  2. Direct extubation: participants will be extubated immediately after spontaneous breathing trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Reconnection to mechanical ventilation for 1 hour (Experimental): As soon as the success of the spontaneous breathing trial is confirmed, the participant will be kept on the mechanical ventilator for 1 hour using the previous ventilatory parameters and, afterwards, extubated.
  Interventions: Other: Reconnection to mechanical ventilation for 1 hour
- Direct extubation (Active Comparator): The participant will be extubated immediately after the spontaneous breathing trial.
  Interventions: Other: Direct extubation

INTERVENTIONS:
Other: Reconnection to mechanical ventilation for 1 hour — As soon as the success of the spontaneous breathing trial is confirmed, the participant will be kept on the mechanical ventilator for 1 hour using the previous ventilatory parameters and, afterwards, extubated.
  Arms: Reconnection to mechanical ventilation for 1 hour
Other: Direct extubation — The participant will be extubated immediately after the spontaneous breathing trial.
  Arms: Direct extubation

SUMMARY:
The aim of this study is to evaluate the feasibility to perform a future larger clinical trial to analyze whether the mechanical ventilation reconnection for 1 hour after a successful spontaneous breathing trial reduces the risk of reintubation or death at 7 days in participants with more than 72 hours of mechanical ventilation. The study will compare two weaning strategies in critically ill participants admitted to intensive care units, with more than 72 hours of mechanical ventilation and with a successful spontaneous breathing trial:

1. Reconnection to mechanical ventilation for 1 hour followed by extubation;
2. Direct extubation.

Follow-up will be until hospital discharge or death.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years;
* Admission to the intensive care unit;
* Orotracheal intubation;
* Mechanical ventilation for more than 72 hours;
* Spontaneous breathing trial (according to the study protocol) successful and considered able to be extubated.

Exclusion Criteria:

* Patients unable to obey commands;
* Unplanned extubation;
* Neuromuscular disease and cervical spinal cord injury;
* Tracheostomy;
* Contraindication for cardiopulmonary resuscitation or reintubation;
* Absence of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-11-02 (Actual); Primary Completion 2024-03-22 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
Feasibility to complete the study according to the planned schedule and with adherence above 90% to the procedures of the experimental and control groups | At day of extubation
  Defined as the capability to complete the study according to the planned schedule and with adherence above 90% to the procedures of the experimental group (mechanical ventilation reconnection for 1 hour [+/-10 min] after spontaneous breathing trial followed by extubation) and control (extubation immediately after spontaneous breathing trial).

SECONDARY OUTCOMES:
Extubation failure within 7 days | Up to 7 days after extubation
  Defined as a composite criterion of reintubation or death 7 days after extubation; Weaning failure will be defined as failure within 7 days after extubation requiring reintubation and invasive mechanical ventilation, whether post-extubation noninvasive ventilation was used or not. The choice of the composite outcome was made to consider possible participants who die before 7 days without being reintubated.
  The choice of time for the 7-day outcome was based on the fact that the time interval to define extubation success varies in the literature, and on the evidence that many participants are reintubated after 48-72 hours, making these times early to assess reintubation, especially in cases of prophylactic use of noninvasive ventilation or post-extubation high flow nasal cannula.
Ventilator-free days in 28 days | Up to 28 days after randomization
  Defined as the number of days from the time of extubation and initiation of unassisted breathing to day 28 after randomization. If a participant dies before day 28, days without ventilation will be counted as zero. If a participant is reintubated and returned to mechanical ventilation and is later extubated again and remains on unassisted breathing through day 28, ventilation-free days will be counted from the end of the last assisted breathing period through day 28. One period of invasive mechanical ventilation lasting less than 24 hours and for the purposes of the surgical procedure will count as 1 day free of mechanical ventilation. Participants who are discharged from the hospital on unassisted breathing before 28 days will be considered ventilator-free for the remaining days up to 28 days.
Length of stay in the intensive care unit | At ICU discharge, up to 90 days
  Length of hospital stay from randomization to intensive care unit discharge
Length of hospital stay | At hospital discharge, up to 90 days
  Length of hospital stay from randomization to hospital discharge
Mortality in the intensive care unit | At intensive care unit discharge, up to 90 days
  Mortality from randomization to intensive care unit discharge
Hospital mortality | At hospital discharge, up to 90 days
  Mortality from randomization to hospital discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Hospitalar Unimed de Joinville, Joinville, Santa Catarina, Brazil

IPD SHARING:
Plan to Share IPD: No
Data will be made available after reasonable request and it has been discussed among the steering committee